CLINICAL TRIAL: NCT05686005
Title: The Efficacy of Oral Versus Intravenous Tranexamic Acid in Functional Endoscopic Sinus Surgery. A Prospective, Randomized, Double-blind Controlled Trial.
Brief Title: Tranexamic Acid in Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Samir Abdelsalam, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 237/ 2022
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Oral tranexamic (Active Comparator): The participants will receive 4 tablets of tranexamic acid 500mg (equal 2gm) 2 hours before surgery in the ward.
  Interventions: Drug: Oral tranexamic acid
- Intravenous tranexamic (Active Comparator): The participants will receive 15 mg/kg in a 20ml syringe slowly tranexamic acid during induction.
  Interventions: Drug: Intravenous tranexamic acid

INTERVENTIONS:
Drug: Oral tranexamic acid — 4 tablets of tranexamic acid 500mg (equal 2gm) 2 hours before surgery in the ward.
  Arms: Oral tranexamic
Drug: Intravenous tranexamic acid — 15mg/kg of tranexamic acid in a 20ml syringe slowly intravenous during induction.
  Arms: Intravenous tranexamic

SUMMARY:
The purpose of the study is to compare the effect of oral tranexamic acid vs. intravenous in decreasing bleeding and improving the field during FESS.

DETAILED DESCRIPTION:
The use of tranexamic acid during Intraoperative bleeding in functional endoscopic sinus surgery (FESS) improves the outcome. Bleeding is one of the most devastating complications during fess. Tranexamic acid is used in open heart surgery to improve the surgical field.

Using oral vs. intravenous forms of the drug will add to our knowledge and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I or II.
* Sex: Both sexes.
* Age between 18 and 40 years.
* Patients scheduled for FESS under general anesthesia.

Exclusion Criteria:

* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* History of venous or arterial thrombosis.
* history of cardiovascular diseases including AF, IHD, or hypertension.
* History of chest problems including pulmonary embolism, bronchial asthma and COPD.
* History of cerebrovascular stroke.
* History of drug or alcohol abuse.
* Taking opioids or sedative medications.
* Hepatic or renal failure.
* Bleeding disorders, antiplatelets (aspirin, clopidogrel) or anticoagulant (warfarin).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative field bleeding | At 30 minutes after surgery start
  The Wormald grading system for bleeding during endoscopic sinus surgery (0= no bleeding and 10= severe bleeding with sphenoid fills < 10 seconds)

SECONDARY OUTCOMES:
Incidence of the common adverse effects | At 24 hours
  Postoperative nasal bleeding, nausea, and vomiting.
Post operative D-dimer | At 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Ain Shams University, Cairo, Egypt